CLINICAL TRIAL: NCT02623101
Title: In Vivo Reflectance Confocal Microscopy, a Novel Non-invasive Tool for Diagnosing Skin Cancer - A Randomized Controlled Trial
Brief Title: Reflectance Confocal Microscopy in Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Mavig GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RCM-onco ZonMw-1
Record Dates: First submitted 2015-11-10; First posted 2015-12-07 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Basal Cell
Keywords: Reflectance confocal microscopy; Basal cell carcinoma; Biopsy; Diagnostics
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Microscopy, Confocal; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care procedure (Active Comparator): Clinical suspected basal cell carcinomas, of all subtypes, will be diagnosed by conventional 3mm punch biopsy of the most clinical suspicious part of the lesion. Punch biopsies will be performed under local anesthetics using 1% xylocaine/adrenaline. Hematoxylin/eosin stained sections of the punch biopsies will be evaluated by an experienced pathologist. Subjects will receive surgical excision according to subtype.
  When there is any doubt by reflectance confocal microscopic diagnosis, a punch biopsy will also be obtained and the lesion will be excized when the biopsy reveals a basal cell carcinoma.
  Interventions: Procedure: Punch biopsy; Procedure: Surgical excision
- Reflectance confocal microscopy (RCM) (Experimental): The Vivascope 1500 and Vivascope 3000 (handheld divice) will be used (CE certified, Lucid Technologies, Henrietta, NY, USA). Reflectance confocal microscopy (RCM) imaging will be performed on clinical suspected basal cell carcinomas, of all subtypes. When there are signs of a basal cell carcinoma imaged by RCM, subjects will receive surgical excision according to subtype. When there is any doubt by RCM diagnosis, a punch biopsy will also be obtained and the lesion will be excized when the biopsy reveals a basal cell carcinoma.
  Interventions: Device: Reflectance confocal microscopy; Procedure: Surgical excision

INTERVENTIONS:
Device: Reflectance confocal microscopy — Non-invasive imaging of the lesion
  Other Names: Confocal microscopy; Vivascope 1500; Vivascope 3000
  Arms: Reflectance confocal microscopy (RCM)
Procedure: Punch biopsy — Obtaining a skin sample of the suspicious lesion under local anesthetics
  Other Names: Biopsy
  Arms: Standard of care procedure
Procedure: Surgical excision — Excision of the basal cell carcinoma lesion under local anesthetics
  Other Names: Surgical removal; Surgery

SUMMARY:
Skin cancer is the most common cancer and its incidence is increasing rapidly. The rising number of skin cancer may result in long waiting lists for consultation at departments for dermatological care and in increasing health care costs. In case of suspicion on skin cancer it is of utmost importance to diagnose and treat in an early phase, preferable in a patient friendly manner. Skin cancer comprises melanoma and non-melanoma skin cancer (NMSC: basal cell carcinoma (BCC), squamous cell carcinoma (SCC) and its precursors actinic keratosis (AK) and Bowen disease). As BCC is the most common skin cancer type with an estimated incidence of 51,000 new tumors in 2015 (The Netherlands), this study will focus on this skin cancer type. In case of suspicion on BCC, at present, the pathological examination of a biopsy is the gold standard for diagnosing a BCC. With the implementation of non invasive diagnosis by reflectance confocal microscopy (RCM) in routine patient care settings the diagnosis can be assessed at the first consultation in a non-invasive way and the patient can be treated instantly.

Overall, the aim of this study is to investigate whether reflectance confocal microscopy can correctly identify the subtype of basal cell carcinoma.

Study design: Randomized controlled trail. Comparison with usual care: punch biopsy and excision.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE:

Skin cancer is the most common cancer and its incidence is increasing rapidly in Western countries. In the Netherlands the registry of skin cancer is poor, however based on recent literature and guidelines the investigators estimate the number of new malignant skin tumors and the precursor actinic keratosis (AK) in 2015 at around 235,278, having a major impact on the health care system. Moreover, it is predicted that numbers of skin cancer will rise with 4.5-8% per year, depending on the type of skin cancer. Skin cancer comprises melanoma and non-melanoma skin cancer (NMSC: basal cell carcinoma (BCC), squamous cell carcinoma (SCC) and its precursors actinic keratosis (AK) and Bowen disease). In case of suspicion on NMSC, at present, the pathological examination of a biopsy is the gold standard. In case of clinical suspicion on AK, the diagnosis is made à vue, without pathological confirmation. In the United States, already in 2003, skin cancer was found to be among the most costly of all cancers to treat, thus, it is evident that skin cancer places an enormous burden on western healthcare systems with increasing costs. As BCC is the most common skin cancer (about 75% of all skin cancers) with an estimated incidence of 51,000 new tumors in 2015, this study will focus on this skin cancer type.

HEALTH CARE EFFICIENCY PROBLEM:

As described above, the incidences of the various malignant skin tumours are increasing dramatically. The rising number of skin cancer may result in long waiting lists for consultation at departments for dermatological care and in increasing health care costs. In case of suspicion on skin cancer it is of utmost importance to diagnose and treat in an early phase, preferable in a patient friendly manner. With the implementation of reflectance confocal microscopy (RCM) in routine patient care settings the diagnosis is assessed at the first consultation and the patient can be treated instantly. A second consultation for explaining the diagnosis is than not necessary, which time can then be used for other new patients. Also, with the conventional diagnostic procedure (pathological investigation of a skin biopsy) the investigators experience in 29% of the cases a sample error, so the BCC subtype is not correctly identified, and as treatment depends on BCC subtype many patients need a subsequent treatment because of treatment failure or recurrence. Also for pathologists, to examine skin tumor after skin tumor is not that efficient and challenging. More pathologists are needed if there will not be other diagnostic techniques in the future. RCM will also, not unimportantly, lower the costs for diagnosing skin cancer.

USUAL CARE:

Currently, in case of suspicion on NMSC, including BCC, an invasive diagnostic biopsy for pathological examination is performed.Treatment choices depend on BCC subtype.

THE INTERVENTION TO BE INVESTIGATED:

RCM is a non-invasive imaging technique. It provides real time images of cell- and tissue structures and dynamics in situ, without the need for ex vivo tissue samples. RCM visualizes human skin up to a depth of around 250 μm. Most, but not all tumors can be visualized. For thicker tumors RCM may help to find the optimal localization to perform a biopsy, as superficial features in these tumors may help to spot these. Moreover, the whole tumor can be imaged by RCM and a diagnosis can be made instantly.

RCM features for skin cancer are reported, which showed a high correlation with conventional pathological features. These features allow to diagnose AK and SCC, and subtypes in BCC (superficial, nodular, micronodular, infiltrative and mixed type BCCs).

RCM in the RELEVANCE FOR PRACTICE

Skin cancer is responsible for 50% of the costs in dermatological patient care, 75-80% of these costs are caused by BCC. These costs will increase even more, as incidence rates will rise further. As described above, the gold standard is pathological investigation of a biopsy or of an excision. However, pathological diagnosis of a biopsy often results in sampling errors, as only a small part of the tumor is investigated resulting in potentially inappropriate chosen therapies. The subtypes of BCC are treated differently. As a sample error may lead to treatment failures or recurrences, other subsequent treatments are needed, increasing costs. In addition, the conventional method is unfriendly for patients, as it is invasive, painful, scarring, and the diagnosis is not instantly available. In order to implement patient friendly RCM in daily BCC care, a large prospective study is needed. The ability of RCM in determining the correct diagnosis and subtyping BCC needs to be investigated as well as preparing protocols for use in patient care. It is believed that this diagnostic imaging technique will be more cost-effective and more patient friendly as compared to the biopsy procedure, the gold standard at present. Therefore, the purpose of this study is to investigate whether reflectance confocal microscopy can correctly identify the subtype of basal cell carcinoma.

Study design: Randomized controlled trail. Comparison with usual care; punch biopsy and excision.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to adhere to all requirements of the study
* Patients must be willing to give written informed consent
* Clinically diagnosed/ clinical suspicion of basal cell carcinoma

Exclusion Criteria:

* Participating in other investigational research currently or in the previous 28 days before the study
* Patient is having a medical condition which excludes participating the research, according to the investigator
* Incapacitated subjects will not be included
* Lesion(s) on parts of the body which do not allow to adequately image the tumour with RCM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2015-12-01; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The number of correctly identified basal cell carcinoma and the subtype by Reflectance confocal microscopy validated by histopathological examination of the excision specimen | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Quality of life (Qol) | Through study completion, an average of 3 years
  VAS (Visual analogue scale)
Cost effectiveness of Reflectance confocal microscopy as diagnostic tool to diagnose basal cell carcinoma | Through study completion, an average of 3 years
  Productivity Cost Questionnaire (IMCQ, generic instrument for measuring medical costs)
Quality Adjusted Live Years (QALY's) | Through study completion, an average of 3 years
  EQ-5D-5L health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: M JP Gerritsen, MD, PhD, Principal Investigator — Radboud University Medical Center, Department of Dermatology
Locations (3):
- Netherlands (3):
  - Canisius Wilhelmina Hospital, Nijmegen
  - Radboud University Medical Center, Nijmegen
  - Rijnstate Hospital, Velp

REFERENCES:
- [Background] Flohil SC, de Vries E, Neumann HA, Coebergh JW, Nijsten T. Incidence, prevalence and future trends of primary basal cell carcinoma in the Netherlands. Acta Derm Venereol. 2011 Jan;91(1):24-30. doi: 10.2340/00015555-1009. PMID 21264452
- [Background] Flohil SC, van der Leest RJ, Dowlatshahi EA, Hofman A, de Vries E, Nijsten T. Prevalence of actinic keratosis and its risk factors in the general population: the Rotterdam Study. J Invest Dermatol. 2013 Aug;133(8):1971-8. doi: 10.1038/jid.2013.134. Epub 2013 Mar 19. PMID 23510990
- [Background] Housman TS, Feldman SR, Williford PM, Fleischer AB Jr, Goldman ND, Acostamadiedo JM, Chen GJ. Skin cancer is among the most costly of all cancers to treat for the Medicare population. J Am Acad Dermatol. 2003 Mar;48(3):425-9. doi: 10.1067/mjd.2003.186. PMID 12637924
- [Background] Wolberink EA, Pasch MC, Zeiler M, van Erp PE, Gerritsen MJ. High discordance between punch biopsy and excision in establishing basal cell carcinoma subtype: analysis of 500 cases. J Eur Acad Dermatol Venereol. 2013 Aug;27(8):985-9. doi: 10.1111/j.1468-3083.2012.04628.x. Epub 2012 Jul 3. PMID 22759209
- [Background] Peppelman M, Wolberink EA, Blokx WA, van de Kerkhof PC, van Erp PE, Gerritsen MJ. In vivo diagnosis of basal cell carcinoma subtype by reflectance confocal microscopy. Dermatology. 2013;227(3):255-62. doi: 10.1159/000354762. Epub 2013 Oct 18. PMID 24158236
- [Background] Peppelman M, Wolberink EA, Koopman RJ, van Erp PE, Gerritsen MJ. In vivo Reflectance Confocal Microscopy: A Useful Tool to Select the Location of a Punch Biopsy in a Large, Clinically Indistinctive Lesion. Case Rep Dermatol. 2013 Apr 25;5(1):129-32. doi: 10.1159/000351258. Print 2013 Jan. PMID 23687492
- [Background] Peppelman M, Nguyen KP, Hoogedoorn L, van Erp PE, Gerritsen MJ. Reflectance confocal microscopy: non-invasive distinction between actinic keratosis and squamous cell carcinoma. J Eur Acad Dermatol Venereol. 2015 Jul;29(7):1302-9. doi: 10.1111/jdv.12806. Epub 2014 Oct 30. PMID 25357235
- [Background] Hoogedoorn L, Peppelman M, Blokx WAM, van Erp PEJ, Gerritsen MP. Prospective differentiation of clinically difficult to distinguish nodular basal cell carcinomas and intradermal nevi by non-invasive Reflectance Confocal Microscopy: a case series study. J Eur Acad Dermatol Venereol. 2015 Feb;29(2):330-336. doi: 10.1111/jdv.12548. Epub 2014 May 20. PMID 24841762
- [Background] Longo C, Lallas A, Kyrgidis A, Rabinovitz H, Moscarella E, Ciardo S, Zalaudek I, Oliviero M, Losi A, Gonzalez S, Guitera P, Piana S, Argenziano G, Pellacani G. Classifying distinct basal cell carcinoma subtype by means of dermatoscopy and reflectance confocal microscopy. J Am Acad Dermatol. 2014 Oct;71(4):716-724.e1. doi: 10.1016/j.jaad.2014.04.067. Epub 2014 Jun 11. PMID 24928707
- [Derived] Peppelman M, Nguyen KP, Alkemade HA, Maessen-Visch B, Hendriks JC, van Erp PE, Adang EM, Gerritsen MJ. Diagnosis of Basal Cell Carcinoma by Reflectance Confocal Microscopy: Study Design and Protocol of a Randomized Controlled Multicenter Trial. JMIR Res Protoc. 2016 Jun 30;5(2):e114. doi: 10.2196/resprot.5757. PMID 27363577